CLINICAL TRIAL: NCT03737643
Title: A Phase III Randomised, Double-Blind, Placebo-Controlled, Multicentre Study of Durvalumab in Combination With Chemotherapy and Bevacizumab, Followed by Maintenance Durvalumab, Bevacizumab and Olaparib in Newly Diagnosed Advanced Ovarian Cancer Patients (DUO-O).
Brief Title: Durvalumab Treatment in Combination With Chemotherapy and Bevacizumab, Followed by Maintenance Durvalumab, Bevacizumab and Olaparib Treatment in Advanced Ovarian Cancer Patients
Acronym: DUO-O
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other); GOG Foundation, Inc. (GOG Foundation) (Unknown); Myriad Genetic Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D081RC00001; 2017-004632-11 (EudraCT Number)
Record Dates: First submitted 2018-10-15; First posted 2018-11-09 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Advanced Ovarian Cancer
Keywords: Advanced Ovarian Cancer; Ovarian neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab; durvalumab; olaparib; CP protocol

STUDY DESIGN:
Intervention Model Description: The study consists of 2 independent cohorts: 3 double-blind treatment arms cohort for patients with no tBRCA mutation, and a single open label arm cohort for patients with tBRCA mutation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Arm 1 (Active Comparator): Platinum-based chemotherapy in combination with bevacizumab and durvalumab placebo (saline IV infusion) followed by maintenance bevacizumab, durvalumab placebo (saline IV infusion) and olaparib placebo (tablets).
  Interventions: Drug: Bevacizumab; Drug: Placebo olaparib; Drug: Durvalumab placebo; Drug: Carboplatin+Paclitaxel
- Arm 2 (Experimental): Platinum-based chemotherapy in combination with bevacizumab and durvalumab followed by maintenance bevacizumab, durvalumab and olaparib placebo.
  Interventions: Drug: Bevacizumab; Drug: Durvalumab; Drug: Placebo olaparib; Drug: Carboplatin+Paclitaxel
- Arm 3 (Experimental): Platinum-based chemotherapy in combination with bevacizumab and durvalumab followed by maintenance bevacizumab, durvalumab and olaparib.
  Interventions: Drug: Bevacizumab; Drug: Durvalumab; Drug: Olaparib; Drug: Carboplatin+Paclitaxel
- tBRCAm cohort (Experimental): Platinum-based chemotherapy in combination with bevacizumab and durvalumab followed by maintenance bevacizumab, durvalumab and olaparib. Bevacizumab is optional according to local practice.
  Interventions: Drug: Bevacizumab; Drug: Durvalumab; Drug: Olaparib; Drug: Carboplatin+Paclitaxel

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab by intravenous infusion. In tBRCAm cohort bevacizumab is optional according to local practice.
Drug: Durvalumab — Durvalumab by intravenous infusion
  Arms: Arm 2; Arm 3; tBRCAm cohort
Drug: Olaparib — Olaparib tablets
  Arms: Arm 3; tBRCAm cohort
Drug: Placebo olaparib — Placebo tablets to match olaparib
  Arms: Arm 1; Arm 2
Drug: Durvalumab placebo — Matching placebo for intravenous infusion
  Arms: Arm 1
Drug: Carboplatin+Paclitaxel — Standard of care chemotherapy

SUMMARY:
This is a Phase III randomised, double-blind, multi-centre study to evaluate the efficacy and safety of durvalumab in combination with standard of care platinum based chemotherapy and bevacizumab followed by maintenance durvalumab and bevacizumab or durvalumab, bevacizumab and olaparib in patients with newly diagnosed advanced ovarian cancer.

DETAILED DESCRIPTION:
Eligible patients will be those patients with newly diagnosed, histologically confirmed advanced (Fédération Internationale de Gynécologie et d'Obstétrique [FIGO] Stage III-IV) ovarian, primary peritoneal cancer and/or fallopian-tube cancer. All patients should be candidates for cytoreductive surgery which could be conducted as immediate upfront primary surgery following diagnosis or can be conducted after initiation of platinum based neoadjuvant chemotherapy. All patients should be eligible to start first line platinum based chemotherapy in combination with bevacizumab.

The study aims to evaluate the efficacy and safety of standard of care (SoC) platinum-based chemotherapy and bevacizumab followed by maintenance bevacizumab either as monotherapy, or in combination with durvalumab, or in combination with durvalumab and olaparib. Therefore, this study aims to see which combination allows patients to live longer without the cancer coming back or getting worse. The study is also looking to see which combination makes patients live longer and how the treatment and the cancer affects their quality of life.

ELIGIBILITY:
Key Inclusion Criteria:

Female patients with newly diagnosed, histologically confirmed, advanced (Stage III-IV) high grade epithelial ovarian cancer including high grade serious, high grade endometriod, clear cell ovarian cancer or carcinosarcoma, primary peritoneal cancer and / or fallopian-tube cancer

* Patients must be aged ≥18 years of age. For patients enrolled in Japan that are aged <20 year
* All patients should be candidates for cytoreductive surgery either: upfront primary surgery OR plan to undergo chemotherapy with interval debulking surgery
* Evidence of presence or absence of BRCA1/2 mutation in tumour tissue
* Mandatory provision of tumour sample for centralised tBRCA testing
* ECOG performance status 0-1
* Patients must have preserved organ and bone marrow function
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test

Key Exclusion Criteria:

Non-epithelial ovarian cancer, borderline tumors, low grade epithelial tumors or mucinous histology

* Prior systemic anti-cancer therapy for ovarian cancer
* Inability to determine the presence or absence of a deleterious or suspected deleterious BRCA mutation
* Prior treatment with PARP inhibitor or immune mediated therapy
* Planned intraperitoneal cytotoxic chemotherapy
* Active or prior documented autoimmune or inflammatory disorders
* Patients considered a poor medical risk due to a serious, uncontrolled intercurrent illness
* Clinically significant cardiovascular disease
* Patients with known brain metastases
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of study treatment and of low potential risk for recurrence (patients who have received prior adjuvant chemotherapy for early stage breast cancer may be eligible, provided that it was completed ≥3 years prior to registration, and that the patient remains free of recurrent or metastatic disease)
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
  * Endometrial cancer FIGO Stage IA, Grade 1 or Grade 2
* Persistent toxicities CTCAE Grade >2 caused by previous cancer therapy
* Patients with a known hypersensitivity to olaparib, durvalumab or any of the excipients of these products and to the combination/comparator agents
* Breast feeding women

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All female patients newly diagnosed with advanced ovarian cancer
Enrollment: 1407 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2025-03-28 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) - in non-tBRCA HRD positive patients | Approximately 4 years
  Defined as time from randomisation to first progression by investigator assessment using modified RECIST 1.1 or death (by any cause in the absence of progression)
Progression Free Survival (PFS) - in all non-tBRCA patients | Approximately 4 years
  Defined as time from randomisation to first progression by investigator assessment using modified RECIST 1.1 or death (by any cause in the absence of progression)

SECONDARY OUTCOMES:
Progression Free Survival (PFS) - in non-tBRCAm patients | Approximately 4 years
  Defined as time from randomisation to first progression by investigator assessment using modified RECIST 1.1 or death (by any cause in the absence of progression)
Overall Survival (OS) - in non-tBRCA HRD positive patients and in all non-tBRCA patients | Approximately 7 years
  Defined as the time from randomisation to death due to any cause
Second Progression (PFS2) - in non-tBRCAm patients | Approximately 7 years
  Defined as time from randomisation to second progression by investigator assessment of radiological progression, symptomatic progression or death (by any cause in the absence of progression)
Health-related quality of life - in non-tBRCAm patients | Approximately 4 years
  Change from baseline in the physical functioning subscale of the EORTC-QLQ-C30
Pathological Complete Response (pCR) - in non-tBRCAm patients | Approximately 4 years
  Defined as the proportion of patients with pCR in patients undergoing IDS
The pharmacokinetics (PK) and immunogenicity of durvalumab and olaparib as determined by peak concentration - in non-tBRCAm patients | Approximately 4 years
  Determination of durvalumab concentration in serum and olaparib concentration in plasma in a subset of patients
Objective Response Rate (ORR) - in non-tBRCAm patients | Approximately 4 years
  Defined as the number (%) of patients with at least one investigator-assessed visit response of CR or PR as per RECIST 1.1
Duration of response (DoR) - in non-tBRCAm patients | Approximately 4 years
  Defined as the time form the date of first documented response (CR/PR) until the first progression or death in the absence of disease progression
Time to first subsequent therapy (TFST) - in non-tBRCAm patients | Approximately 7 years
  Time elapsed from randomisation to first subsequent therapy or death
Time to second subsequent therapy (TSST) - in non-tBRCAm patients | Approximately 7 years
  Time elapsed from randomisation to second subsequent therapy or death
Time to discontinuation or death (TDT) - in non-tBRCAm patients | Approximately 4 years
  Time elapsed from randomisation to study treatment discontinuation or death
PFS - in tBRCAm patients | Approximately 4 years
  To assess the potential additional clinical benefit of durvalumab added to SoC and olaparib in the first line treatment of tBRCAm patients
PFS2 - in tBRCAm patients | Approximately 7 years
  To assess the potential additional clinical benefit of durvalumab added to SoC and olaparib in the first line treatment of tBRCAm patients
ORR - in tBRCAm patients | Approximately 4 years
  To assess the potential additional clinical benefit of durvalumab added to SoC and olaparib in the first line treatment of tBRCAm patients
ORR pre-surgery in IDS group - in tBRCAm patients | Approximately 4 years
  To assess the potential additional clinical benefit of durvalumab added to SoC and olaparib in the first line treatment of tBRCAm patients
Duration of response (DoR) - in tBRCAm patients | Approximately 4 years
  To assess the potential additional clinical benefit of durvalumab added to SoC and olaparib in the first line treatment of tBRCAm patients
Time to first subsequent therapy (TFST) - in tBRCAm patients | Approximately 7 years
  To assess the potential additional clinical benefit of durvalumab added to SoC and olaparib in the first line treatment of tBRCAm patients
Time to second subsequent therapy (TSST) - in tBRCAm patients | Approximately 7 years
  To assess the potential additional clinical benefit of durvalumab added to SoC and olaparib in the first line treatment of tBRCAm patients
Time to discontinuation or death (TDT) - in tBRCAm patients | Approximately 4 years
  To assess the potential additional clinical benefit of durvalumab added to SoC and olaparib in the first line treatment of tBRCAm patients
Health-related quality of life - in tBRCAm patients | Approximately 4 years
  Change from baseline in the physical functioning subscale of the EORTC-QLQ-C30
Proportion of patients with pCR in patients undergoing IDS - in tBRCAm patients | Approximately 4 years
  To assess the potential additional clinical benefit of durvalumab added to SoC and olaparib in the first line treatment of tBRCAm patients

OTHER OUTCOMES:
Safety and tolerability of drugs by assessment of AEs/SAEs | Approximately 4 years
  Graded according to the National Cancer Institute (NCI CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Harter, Principal Investigator — European Network of Gynaecological Oncological Trial Groups (ENGOT); Carol Aghajanian, Principal Investigator — GOG
Locations (181):
- United States (25):
  - Research Site, Foothill Ranch, California
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, San Francisco, California
  - Research Site, Tampa, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Hinsdale, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Towson, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Springfield, Missouri
  - Research Site, Middletown, New Jersey
  - Research Site, Montvale, New Jersey
  - Research Site, Albany, New York
  - Research Site, New York, New York
  - Research Site, Uniondale, New York
  - Research Site, Durham, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Hilliard, Ohio
  - Research Site, Tulsa, Oklahoma
  - Research Site, Lancaster, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Salt Lake City, Utah
- Austria (4):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Vienna
- Belgium (5):
  - Research Site, Aalst
  - Research Site, Leuven
  - Research Site, Namur
  - Research Site, Ostend
  - Research Site, Sint-Niklaas
- Brazil (7):
  - Research Site, Barretos
  - Research Site, Florianópolis
  - Research Site, Fortaleza
  - Research Site, Londrina
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Bulgaria (4):
  - Research Site, Burgas
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
- Canada (7):
  - Research Site, Calgary, Alberta
  - Research Site, Barrie, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Rimouski, Quebec
- China (24):
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Dalian
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Jinhua
  - Research Site, Kunming
  - Research Site, Lanzhou
  - Research Site, Luzhou
  - Research Site, Nanchong
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Nantong
  - Research Site, Shanghai
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhengzhou
  - Research Site, Zhuhai
- Denmark (5):
  - Research Site, Aalborg
  - Research Site, Aarhus N
  - Research Site, Odense
  - Research Site, Roskilde
  - Research Site, Vejle
- Finland (3):
  - Research Site, Kuopio
  - Research Site, Oulu
  - Research Site, Turku
- France (9):
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Limoges
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Saint-Herblain
  - Research Site, Vandœuvre-lès-Nancy
- Germany (36):
  - Research Site, Bad Homburg
  - Research Site, Berlin
  - Research Site, Bielefeld
  - Research Site, Bonn
  - Research Site, Brandenburg
  - Research Site, Cologne
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Essen
  - Research Site, Esslingen am Neckar
  - Research Site, Frankfurt
  - Research Site, Freiburg im Breisgau
  - Research Site, Fürth
  - Research Site, Greifswald
  - Research Site, Gütersloh
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Jena
  - Research Site, Karlsruhe
  - Research Site, Kassel
  - Research Site, Kiel
  - Research Site, Leipzig
  - Research Site, Ludwigsburg
  - Research Site, Lübeck
  - Research Site, Mainz
  - Research Site, Mannheim
  - Research Site, München
  - Research Site, Offenbach
  - Research Site, Oldenburg
  - Research Site, Rosenheim
  - Research Site, Rostock
  - Research Site, Saalfeld
  - Research Site, Schweinfurt
  - Research Site, Tübingen
  - Research Site, Ulm
  - Research Site, Worms
- Hungary (6):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Kaposvár
  - Research Site, Szeged
  - Research Site, Zalaegerszeg
- Italy (10):
  - Research Site, Brescia
  - Research Site, Lecce
  - Research Site, Lecco
  - Research Site, Milan
  - Research Site, Mirano
  - Research Site, Napoli
  - Research Site, Reggio Calabria
  - Research Site, Reggio Emilia
  - Research Site, Roma
  - Research Site, Torino
- Japan (15):
  - Research Site, Fukuoka
  - Research Site, Kashiwa-shi
  - Research Site, Kobe
  - Research Site, Kōtoku
  - Research Site, Kurume-shi
  - Research Site, Kyoto
  - Research Site, Minatoku
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Okayama
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
  - Research Site, Sunto-gun
  - Research Site, Toyoake-shi
- Peru (4):
  - Research Site, Bellavista
  - Research Site, La Libertad
  - Research Site, Lima
  - Research Site, San Isidro
- Poland (4):
  - Research Site, Gdynia
  - Research Site, Lodz
  - Research Site, Szczecin
  - Research Site, Warsaw
- Research Site, Floreşti, Romania
- South Korea (4):
  - Research Site, Goyang-si
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (4):
  - Research Site, Córdoba
  - Research Site, Madrid
  - Research Site, Terrassa(Barcelona)
  - Research Site, Vigo
- Turkey (Türkiye) (4):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961